CLINICAL TRIAL: NCT04251832
Title: Efficacy of Sodium Thiosulfate in Shoulder Pain in Calcific Tendinitis of the Rotator Cuff
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soraia Azevedo (Other)
Responsible Party: Sponsor-Investigator, Soraia Azevedo, Principal Investigator, Unidade Local de Saúde do Alto Minho
Organization: Unidade Local de Saúde do Alto Minho (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STShoulderPain
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Sodium Thiosulfate; Calcific Tendinitis; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — sodium thiosulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ultrasound guided percutaneous lavage with STS (Experimental): Ultrasound guided percutaneous lavage with a single needle technic. A total of 10 mL of lidocaine 1% will be injected in the subcutaneous tissues, the subacromial bursa and over the surface of the calcific deposit. A 21 G pediatric spinal needle will be used for the procedure to prevent needle clogging by calcific debris. When backflow of calcific material could be identified in the syringe, lavage of the deposit will be performed using sodium thiosulfate 25 %: a volume of 1 mL of sodium thiosulfate will be prepared in a syringe and successive propulsion and aspiration will be performed. The procedure will be repeated until the backflow becomes clear. At the end of the procedure 1 mL (250 mg) of thiosulfate will be injected inside the calcific deposit. Finally, 1.5 mL of methylprednisolone will be injected in the SAB.
  Only a single procedure will be performed and the outcomes measured after 1 week, 1 month and 3 months.
  Interventions: Drug: Sodium Thiosulfate
- Ultrasound guided percutaneous lavage without STS (Active Comparator): Ultrasound guided percutaneous lavage with a single needle technic. A total of 10 mL of lidocaine 1% will be injected in the subcutaneous tissues, the subacromial bursa and over the surface of the calcific deposit. A 21 G pediatric spinal needle will be used for the procedure to prevent needle clogging by calcific debris. When backflow of calcific material could be identified in the syringe, lavage of the deposit will be performed using of saline solution and successive propulsion and aspiration will be performed. The procedure will be repeated until the backflow becomes clear. Finally, 1.5 mL of methylprednisolone will be injected in the SAB.
  Only a single procedure will be performed and the outcomes measured after 1week, 1month and 3months
  Interventions: Drug: Sodium Thiosulfate

INTERVENTIONS:
Drug: Sodium Thiosulfate — Ultrasound guided percutaneous lavage with and without Sodium Thiosulfate

SUMMARY:
Calciﬁc tendinitis of the rotator cuff is one of the most common causes of shoulder pain. Ultrasound guided percutaneous lavage (UGPL or barbotage or irrigation) of calcific tendinopathy is indicated when conservative treatments (physiotherapy, nonsteroidal anti-inflammatory drugs) have failed. Our hypothesis is that lavage followed by intra-calcic injection of STS could fasten the dissolution of the calcific deposit. In view of the short half-life of this molecule the investigators hypothesize that this would happen within the first month after the procedure. Therefore, the investigatorschose to assess our primary objective at 1 month. Few studies have evaluated the short-term radiographic evolution after lavage.

DETAILED DESCRIPTION:
Calciﬁc tendinitis of the rotator cuff is one of the most common causes of shoulder pain. It is characterized by calcium phosphate crystal deposition in the rotator cuff. Its pathogenesis and etiology remains unclear and the mechanisms leading to this pathological mineralization are still largely unknown. This disorder can lead to a chronic pain during daily or professional activities and to a restriction of range of motion. During the disease, spontaneous resorption can occur with migration of apatite crystals into the subacromial bursa causing severe pain and restriction of movement. Factors associated with the development of symptoms are still unclear although the size and presence of a bursitis on imaging have been shown to be associated with pain.

Ultrasound guided percutaneous lavage (UGPL or barbotage or irrigation) of calcific tendinopathy is indicated when conservative treatments (physiotherapy, nonsteroidal anti-inflammatory drugs) have failed. At this stage, extracorporeal shock wave therapy (ESWT) or subacromial corticosteroid injection can also be discussed. However, a recent network meta-analysis has shown that UGPL could be the treatment of choice compared to the other nonsurgical options such as ESWT or SAI. Arthroscopic removal of the calcific deposit is considered as a second line therapy after failure of UGPL or EWST.

Efficacy of UGPL depends on the type of calcification. Calcific deposits can be differentiated in hard calcifications, usually dense on X-Ray with an acoustic shadow on US, and soft calcifications, with more heterogeneous or faint contours without acoustic shadowing. Some studies observed failure only in patients presenting with a dense and homogeneous calcification type A according to the Molé Classification and also showed that outcome after needling and/or ESWT will be worse in case of dense calcifications, with only 30% of success compared to 61% in patients with soft calcification. These failures are most of the time explained by the persistence of the calcific deposit. In line with this, was found a positive correlation between the decrease of the size of the calcification and the pain score over time; as the calcification became smaller, the pain became less intense.

Several approaches are currently used to facilitate the extraction of the calcification. It has been shown that lavage with warm saline heated at 42°C reduced the procedure duration and improved calcification dissolution. Another randomized controlled study recently reported that lavage with a 2 needle approach also shortened the procedure in hard calcification. However, none of these studies showed an impact on the rate of calcification elimination. Other strategies are therefore needed to treat hard calcification of the rotator cuff.

Sodium thiosulfate (STS) (Na2S2O3) is primarily used to prevent and treat cyanide poisoning. Intravenous STS is also used off-label to treat calciphylaxis leading to a significant decrease of soft-tissue and vascular calcifications. However, its systemic use may be limited by adverse effects, such as gastrointestinal upset, metabolic acidosis, and sodium overload. Thus, alternative local approaches have been developed. Recent reports have shown the interest of topical STS in the treatment of calciphylaxis, tumoral calcinosis associated with connective tissue disease, pseudohypoparathyroidism or hyperphosphatemic familial tumoral calcinosis. For instance, a daily application of topical STS on the calcific lesions of patients with hyperphosphatemic familial tumoral calcinosis led to their decrease after 5 months of treatment. Topical application of STS has also showed an anti-inflammatory effect in patients with calcinosis cutis secondary to connective tissue disease and radiodermatitis. Because deeper calcific deposits are unlikely to be reached by topical therapeutic agents, some authors performed intralesional STS injections in patients with localized cutaneous calciphylaxis. They observed a complete healing of ulcers and remission of disease with only transient localized discomfort during injection. Despite these promising results, the exact mechanisms by which STS is able to dissolve ectopic calcifications remain still unclear.

Recently one study showed that STS was well tolerated with no side effect occurring during ultrasound-guided percutaneous lavage of calcific tendinopathy.

These preliminary results prompted us to study the interest of STS in the treatment of calcific tendinitis. As dense calcifications are associated with higher risk of failure of UGPL, the investigators will select patients to perform a lavage followed by an intralesional injection of STS. The objective of our study is to evaluate the efficacy of sodium thiosulfate lavage in the treatment of shoulder pain in calcific tendinitis. the investigators will also assess its effect on clinical symptoms and radiographic evolution of the calcific deposit and hypothesize that sodium thiosulfate would be well-tolerated and fastened the elimination of the calcific deposit in patients with dense calcifications.

METHODS The current study is a prospective, monocentric, phase II, single group, open label study.

Study population The investigators will include patients referred to the rheumatology department for the treatment of a shoulder pain calcific tendinitis. Inclusion criteria are the following: age over 18 years old; pain for more than 3 months; worsening of symptoms with activities above shoulder level; minimum one the 3 following impingement positive clinical tests (Yocum, Hawkins, Neer); calcification > 5 mm in size on the standard anteroposterior (AP) radiographs. Only type A calcification according the Molé Classification will be included. The exclusion criteria will be: allergy to sodium metabisulfite, asthma, chronic renal disease (creatinine clearance <30 ml/min), Type B or C calcification according the Molé Classification, other shoulder disease (glenohumeral or acromioclavicular osteoarthritis, rotator cuff tear, rheumatoid arthritis); previous percutaneous irrigation of the same calcification.

Baseline clinical, radiological and ultrasonographic evaluation The investigators will recorde the main demographic characteristics: medical history, occupation, dominant hand, presence of nocturnal pain, and day off-work because of the shoulder pain. VAS pain at rest and during activities, shoulder range of motion, DASH score, and EQ5D quality of life VAS score will also be recorded. X-Ray of the affected shoulder will be performed (anteroposterior view in neutral, internal and external rotation and lateral scapula view). Calcifications types will be classified according to Molé at al (A: dense, well defined and circumscribed; B: dense, well-defined and segmented; C: transparent and nonhomogeneous). Surface of the calcification will be measured on the view where the calcification appears the largest. The same view will be used for all measurements during follow-up. Density of the deposit will be evaluated on the same view. All the measurements will be made by an experienced rheumatologist (with 35 years' experience in clinical radiologic evaluation) blinded from the clinical status (ABV).

US evaluation of the affected shoulder will be performed using a GE LogiS8 using a 6-15 MHz linear probe. The investigators will be recorded the maximum size of the calcic deposit in axial and longitudinal view. Calcific shoulder plaques will be classified into 4 types based on their morphology, as previously described. Arc-shaped (an echogenic arc .with clear shadowing); 2. Fragmented or punctate (at least 2 separated echogenic spots or plaques) with shadowing); 3. Fragmented or punctate without shadowing; 4. Nodular (an echogenic nodule without shadowing). Presence of a bursitis (>2 mm thickening of the SAB) and power Doppler signal in and around the calcification will be recorded. For power Doppler imaging, the pulse repetition frequency will be set at 2.4 cm/s and the color gain at the most sensitive level before the appearance of noise. The color flow signal intensity will be graded on a scale of 0 to 3, where 0 represents no signal, 1 = mild (weak, spot-like color flow signal), 2 = moderate (a few rod-like color flow signals), and 3 = severe (multiple rod-like or linear color flow signals).

Intervention All patients will be undergoing a baseline clinical, X-Ray and US evaluation by rheumatologists with 11 years and 5 years' experience in US and US-guided interventions. Patients will be with a US-guided single needle technic. After sterile preparation, local anesthesia will be performed under US guidance. A total of 10 mL of lidocaine 1% will be injected in the subcutaneous tissues, the subacromial bursa and over the surface of the calcific deposit. A 21 G pediatric spinal needle will be used for the procedure to prevent needle clogging by calcific debris. Indeed, introduction of the needle with the stylet prevents the needle to be clogged. Once the needle tip will be inside the calcification, the stylet will be removed, and the lavage could start. When backflow of calcific material could be identified in the syringe, lavage of the deposit will be performed using sodium thiosulfate 25 %: a volume of 1 mL of sodium thiosulfate will be prepared in a syringe and successive propulsion and aspiration will be performed. The procedure will be repeated until the backflow becomes clear. At the end of the procedure 1 mL (250 mg) of thiosulfate will be injected inside the calcific deposit. Finally, 1.5 mL of methylprednisolone will be injected in the SAB.

X-Ray of the shoulder will be performed just after the procedure. Patients will be treated with diclofenac (75 mg LP twice daily) and paracetamol (1000 mg, 4 times a day) for 48 hours then only if needed. Routine use of the shoulder will be allowed without restrictions and all patients had one week off-work.

Follow-up All patients will have follow-up visits at 1 week, 1 month and 3 months after intervention. At each time point, VAS pain at rest and during activities, shoulder range of motion, and DASH score will be recorded. EQ5D quality of life VAS score will be also recorded. X-Ray of the affected shoulder will be performed at each time point and evaluated as previously described. Care will be taken to use the exact same settings (mAs;kV) to allow a proper comparison of the calcific deposit between each evaluation. The evolution of the calcific deposit will be evaluated using a semi-quantitative score as followed: 0: no change or minimal changes; 1: decrease size of the calcification less than 50%; 2: decrease of the calcification between 50 and 90%; 3: more than 90% decrease size or disappearance of the calcification. Surface of the calcification will be measured on the same view than at baseline. US of the affected shoulder will be performed as previously described.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old;
* Pain for more than 3 months;
* Worsening of symptoms with activities above shoulder level;
* Minimum one the 3 following impingement positive clinical tests: Yocum, Hawkins or Neer;
* Calcification > 5 mm in size on the standard anteroposterior radiographs;
* Type A calcification according the Molé Classification .

Exclusion Criteria:

* Allergy to sodium metabisulfite;
* Asthma;
* Chronic renal disease (creatinine clearance <30 ml/min);
* Type B or C calcification according the Molé Classification;
* Other shoulder disease (glenohumeral or acromioclavicular osteoarthritis, rotator cuff tear, rheumatoid arthritis);
* Previous percutaneous irrigation of the same calcification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of the calcific deposit | 1 week, 1 month and 3 months
  Evaluated using a semi-quantitative score as followed: 0: no change or minimal changes; 1: decrease size of the calcification less than 50%; 2: decrease of the calcification between 50 and 90%; 3: more than 90% decrease size or disappearance of the calcification

SECONDARY OUTCOMES:
Visual Analogue Scale pain at rest | 1 week, 1 month and 3 months
  Visual Analogue Scale minimum:"0" - "no pain maximum:"10" - extreme pain
Visual Analogue Scale pain at during activities | 1 week, 1 month and 3 months
  Visual Analogue Scale minimum:"0" - "no pain maximum:"10" - extreme pain
Shoulder range of motion | 1 week, 1 month and 3 months
  Impingement positive clinical tests (Yocum; Hawkins; Neer) Shoulder range of motion
Disabilities of the Arm, Shoulder and Hand score | 1 week, 1 month and 3 months
  Disabilities of the Arm, Shoulder and Hand score: 30 items, scored 1-5; scaled on a 0-100 scale: a higher score indicates greater disability
EuroQol-5D quality of life score | 1 week, 1 month and 3 months
  EuroQol-5D quality of life score, better outcome: 1, worse outcome: -0.4963

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade Local de Saúde do Alto Minho - Hospital Conde de Bertiandos, Ponte de Lima, Portugal